CLINICAL TRIAL: NCT00956098
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Multicenter Trial of Oltipraz for the Evaluation of Efficacy and Safety in the Patients With Liver Fibrosis and Cirrhosis Induced by Chronic Hepatitis Type B or C
Brief Title: Efficacy and Safety of Oltipraz in the Patients With Liver Fibrosis and Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: CJ Cheiljedang Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CJ-OPZ-201 study
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Liver Fibrosis; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — oltipraz

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- oltipraz (Experimental)
  Interventions: Drug: oltipraz

INTERVENTIONS:
Drug: oltipraz — 60mg bid 90mg qd
  Arms: oltipraz
Drug: placebo
  Arms: placebo

SUMMARY:
This study investigated the effectiveness and safety of oltipraz therapy in treating patients with cirrhosis induced by chronic hepatitis type B or C.

DETAILED DESCRIPTION:
Oltipraz [5-(2-pyrazinyl)-4-methyl-1,2-dithiol-3-thione] has been extensively studied as a cancer chemopreventive agent. Comprehensive mechanistic and phase IIa studies supported the notion that oltipraz exerts chemopreventive effects, as supported by Phase IIa human clinical studies of oltipraz on cancer chemoprevention, conducted in Qidong, China. Hepatic stellate cells cause synthesis of large quantities of extracellular matrix. Transforming growth factor beta1 (TGF-beta1), as a key fibrogenic mediator for fibrogenesis after injuries through deposition of extracellular matrix and inhibition of collagenase activity in the liver, is associated with the regulation of cell growth and differentiation and causes synthesis of extracellular matrix proteins and cellular receptors for matrix proteins. Previously, we reported the effectiveness of oltipraz in regeneration of cirrhotic liver, which includes reduction of the intensities of liver fibrotic and cirrhotic nodules, elimination of accumulated extracellular matrix, and regeneration of cirrhotic liver in animal models. Oltipraz completely resolves fibrosis in the cirrhotic liver, thereby improving viability. TGF-beta1 signaling plays an important role in liver fibrogenesis and cirrhosis as evidenced by receptor knockout experiments. No therapeutic agent that is active in interrupting TGF-beta1 signaling is available, proposing that C/EBP serve as a molecular target for the treatment of liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with fibrosis and cirrhosis induced by chronic hepatitis type B or C
* patients with HbsAg, Anti-HCV or HCV RNA positive

Exclusion Criteria:

* treatment with antiviral agents, immunosuppressants, glucocorticoids, within the 6 months or with biphenyl dimethyl dicarboxylate one month
* treatment with any investigational drug (except CJ11555PK or CJ-OPZ-201PK) within one month
* Child-Pugh class C, Use of a mean daily dose of 80 g alcohol with the one month, of enzyme inducers or inhibitors, or of drug abuse that might affect this study
* a known hypersensitivity to oltipraz or its structurally related compounds
* ascites, hemorrhage from varicoses, uncompensated LC with the history of hepatic encephalopathy within the 6 months
* hepatocellular carcinoma (a rising serum level of α-fetoprotein or a suspicious foci on hepatic ultrasonography at screening or), liver transplantation
* pregnancy or lactation, unwillingness of contraception during the study period
* other serious concurrent illness (e.g., severe hemorrhagic GI, renal, pulmonary, neurological, cardiovascular (CHF of class III or above; a history of MI within the past 6 months) diseases, or cancer, autoimmunity or psychological diseases)
* any patients who is inappropriate or has unwillingness of clinical study as judged by participating clinicians
* bilirubin content greater than 2.0 mg/dL, prothrombin time longer than 4 sec, and serum albumin below 2.5 g/dL

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81
Dates: Start 2006-02; Study Completion 2007-02

PRIMARY OUTCOMES:
Ishak fibrosis score | 24 weeks

SECONDARY OUTCOMES:
The Modified Knodell's HAI score | 24 weeks
Child-Pugh score | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - The Catholic University of Korea Holy Family Hospital, Sosa-Dong, Wonmi-Gu, Gyeonggi-do
  - The Catholic University of Korea Seoul St. Mary's Hospital, Banpo-Dong, Seocho-Gu, Seoul